CLINICAL TRIAL: NCT06323525
Title: A Phase 1/2 Single-center Study Evaluating the Safety and Efficacy of TCR Reserved and Power3 (SPPL3) Gene Knock-out Allogeneic CD19-targeting CAR-T Cell (ATHENA-2) Therapy in Adults With Refractory/Relapsed B-cell Lymphoma
Brief Title: TCR Reserved and Power3 (SPPL3) Gene Knock-out Allogeneic CD19-targeting CAR-T Cell Therapy in r/r B Cell Lymphoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, Director of Biotherapeutic Department, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-083
Record Dates: First submitted 2024-03-08; First posted 2024-03-21 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Non-hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — fludarabine; fludarabine phosphate; Injections; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with refractory or relapsed B-cell lymphoma (Experimental): A conditioning chemotherapy regimen of fludarabine and cyclophosphamide will be administered followed by investigational treatment, Power3 (SPPL3) gene knock-out allogeneic CD19-targeting CAR-T.
  Interventions: Biological: TCR reserved and Power3 (SPPL3) gene knock-out allogeneic CD19-targeting CAR-T cell (ATHENA-2 CAR-T); Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: TCR reserved and Power3 (SPPL3) gene knock-out allogeneic CD19-targeting CAR-T cell (ATHENA-2 CAR-T) — Phase 1 dose escalation (3+3): dose 1 (1 × 10^6 cells/kg), dose 2 (3 × 10^6 cells/kg), dose 3 (6 × 10^6 cells/kg); Phase 2: dose of RP2D.
Drug: Fludarabine — Intravenous fludarabine 30~50 mg/m^2/day on days -5, -4, and -3.
  Other Names: Fludarabine Phosphate for Injection
Drug: Cyclophosphamide — Intravenous cyclophosphamide 500~1000 mg/m^2/day on days -5, -4, and -3.
  Other Names: Cyclophosphamide for Injection

SUMMARY:
The safety and efficacy of the chimeric antigen receptor (CAR)-T, a CD19-targeting, TRAC and Power3 (SPPL3) double genes deleted allogeneic CAR-T cell product, are undergoing rigorous evaluation in non-Hodgkin's lymphoma (NHL) subjects from our ATHENA trial (NCT06014073). Unexpectedly, expansion of the initial residual CD3-positive CAR T from products were measured in patients' peripheral blood (PB) without exception. Accompanying with host immune reconstitution and appearance of the detectable B cells, the CD3-positive allogenic CAR T cells exhibited a compelling amplification advantage over CD3-negative CAR T cells. The amplification of CD3-positive CAR T cell population dynamically suppressed host B cell recovery, and presumably surveilled the recurrence or progression of tumors, but did not induce typical Graft-versus-host-disease (GvHD). Additionally, a series of in vitro experiments illustrated that the HLA-mismatched fratricide between host T cells and TCR-reserved Power3 (SPPL3)-deleted allogenic CAR T cells was markedly slashed, which in combination with our observed clinical safety date supported the notion that only genomic deletion of Power3 (SPPL3) gene in allo-CAR T cells is sufficient to overcome GvHD and host T cell-mediated rejection response.

In the ATHENA-2 study, our design is to preserve the expression of the TCR on T cells from healthy donors while selectively disabling the Power3 (SPPL3) gene to prepare ATHENA-2 CAR T cells. This approach harnesses the tonic signaling of CAR T cells, resulting in enhanced persistence and improved response to treatment. The purpose of this study is to evaluate the safety and efficacy of ATHENA-2 in B-cell NHL.

DETAILED DESCRIPTION:
Phase 1 (dose escalation)

In phase 1, 6-18 subjects will be enrolled. Subjects will receive 3 doses of ATHENA-2 CAR-T cell therapy ( 1× 10^6 cells/kg, 3× 10^6 cells/kg, 6 × 10^6 cells/kg) increases from low dose to high dose according to the "3 + 3" principle:

Three (3) subjects are enrolled in a cohort corresponding to a dose level. If 1 subject in a cohort of 3 subjects experiences a dose-limiting toxicity (DLT), 3 additional subjects will be enrolled at the current dose level. For safety purposes, the administration of ATHENA-2 CAR T will be staggered by 28 days between the first two subjects in each cohort. And for each of the remaining cohorts, the administration of ATHENA-2 CAR-T will be staggered by 28 days before enter into the next cohort.

Phase 2 (expansion cohort)

In phase 2, 10 to 12 subjects will be enrolled and receive ATHENA-2 CAR-T cell infusion at dose of recommended phase 2 dose (RP2D), which will be determined based on the maximum tolerated dose (MTD), occurrence of DLT, the obtained efficacy results, pharmacokinetics/pharmacodynamics and other data according to the phase 1.

Objectives:

The primary objectives of the phase 1 are to evaluate the tolerability and safety of ATHENA-2 CAR-T in patients with r/r B-cell NHL, and determine RP2D. The primary purpose of the phase 2 study is to evaluate the efficacy of ATHENA-2 CAR-T in the above population.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 (inclusive).
2. Subjects who meet the following requirements:

   2.1 Histologically confirmed refractory/relapsed B cell NHL, including the following types defined by WHO 2016:
   * Diffuse large B-cell lymphoma not otherwise specified (DLBCL-NOS);
   * Primary mediastinal (thymic) large B-cell lymphoma (PMBCL);
   * Transformed follicular lymphoma (TFL);
   * High-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements (HGBCL);
   * Follicular lymphoma (FL);
   * Mantle cell lymphoma (MCL) (pathologically confirmed, with documentation of monoclonal B cells that have a chromosome translocation t(11;14)(q13;q32) and/or overexpress cyclin D1);
   * Marginal zone lymphoma (MZL), including nodal or splenic marginal zone B-cell lymphoma and mucosa-associated lymphoid tissue (MALT) lymphoma.

   2.2 Relapsed disease is defined as disease progression (PD) after achieving disease remission (including CR and PR) with the latest standard regimen.

   2.3 Refractory disease is defined as no CR to first-line therapy:
   * Evaluation of PD (never reached response or SD) after standard first-line treatment, or
   * SD as best response after at least 4 cycles of first-line therapy (eg,4 cycles of R-CHOP), or
   * PR as best response after at least 6 cycles and biopsy-proven residual disease or disease progression ≤ 6 months of therapy, or
   * Refractory post-autologous stem cell transplant (ASCT): i. Disease progression or relapsed less than or equal to 12 months of ASCT (must have biopsy proven recurrence in relapsed individuals); ii. If salvage therapy is given post-ASCT, the individual must have had no response to or relapsed after the last line of therapy.

   2.4 Individuals who are intolerant to standard treatment can also be included in the study in the investigator's judgment.
3. Individuals must have received adequate prior therapy:

   3.1 For MCL, prior therapy must have included:
   * Anthracycline or bendamustine-containing chemotherapy and
   * Anti-CD20 monoclonal antibody (unless investigator determines that tumor is CD20-negative) and
   * Bruton's tyrosine kinase inhibitor (BTKi).

   3.2 For other types, prior therapy must have included:
   * Anti-CD20 monoclonal antibody (unless investigator determines that tumor is CD20-negative) and
   * Anthracycline containing chemotherapy regimen.

   3.3 For individual with transformed FL must have relapse or refractory disease after transformation to DLBCL.
4. At least 1 measurable lesion: lymph node site with a long axis >1.5cm, extranodal site with a long axis >1.0cm (according to the Lugano2014 criteria). Lesions that have been previously irradiated will be considered measurable only if progression has been documented following completion of radiation therapy.
5. CD19 positive (detected by immunohistochemistry [IHC]).
6. Toxicities due to prior therapy must be stable and recovered to ≤ Grade 1 (except for hematological toxicities and clinically non-significant toxicities such as alopecia).
7. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
8. Absolute neutrophil count (ANC) ≥ 1 x 10^9/L, Platelet count ≥50 x 10^9/L, hemoglobin (Hgb) ≥ 80g/L (hemocytopenia caused by lymphoma invasion of bone marrow is not subject to conditions above).
9. Adequate renal, hepatic, pulmonary and cardiac function defined as:

   9.1 Serum creatinine≤1.5 upper limit of normal (ULN) or creatinine clearance (as estimated by Cockcroft Gault) ≥ 60 mL/min.

   9.2 Serum alanine aminotransferase / aspartate aminotransferase (ALT/AST) ≤ 3 upper limit of normal (ULN); Total bilirubin ≤ 1.5 ULN, except in subjects with 3) Gilbert's syndrome.

   9.3 Cardiac ejection fraction ≥ 50%, no evidence of pericardial effusion as determined by an echocardiogram (ECHO), and no clinically significant electrocardiogram (ECG) findings.

   9.4 Coagulation Function: International Normalized Ratio (INR) ≤ 1.5 times the upper limit of normal (ULN), and Activated Partial Thromboplastin Time (APTT) ≤ 1.5 times ULN.

   9.5 Baseline oxygen saturation >91% on room air.
10. Subjects of both genders who are willing to practice birth control from the time of consent through 6 months after the completion of conditioning chemotherapy. Females of childbearing potential must have a negative serum or urine pregnancy test (females who have undergone surgical sterilization or who have been postmenopausal for at least 2 years are not considered to be of childbearing potential).
11. Voluntarily participate in this clinical trial and sign an informed consent form.

Exclusion Criteria:

1. Expected survival time < 3 months per Principal Investigator's opinion.
2. History of malignancy other than nonmelanoma skin cancer or carcinoma in situ (e.g. cervix, bladder, breast) or follicular lymphoma unless disease free for at least 3 years.
3. Autologous stem cell transplant with therapeutic intent within 3 months of planned ATHENA-2 CAR-T infusion.
4. History of allogeneic stem cell transplantation.
5. Patients who received any immunocellular therapy within 3 months before enrollment.
6. Patients who have used any of the following agents or treatments within a specific period of time:

   6.1 Received any chemotherapy drugs or small molecule targeted drugs within 2 weeks prior to lymphodepletion;

   6.2 Received any monoclonal antibodies, antibody drug conjugates (ADCs), or bispecific antibodies within 3 weeks prior to lymphodepletion;

   6.3 Received radiotherapy within 6 weeks prior to lymphodepletion. However, if disease progressed at the site of radiotherapy, or if there are positive lesions detected by PET-CT at non-radiotherapy sites, enrollment is allowed.
7. Subjects with detectable cerebrospinal fluid malignant cells, or brain metastases, or with a history of central nervous system (CNS) lymphoma or primary CNS lymphoma.
8. Presence of donor-specific anti-HLA antibodies directed against ATHENA-2 CAR-T.
9. History of severe, immediate hypersensitivity reaction attributed to lymphodepletion drugs or any component of ATHENA-2 CAR-T.
10. Presence or suspicion of fungal, bacterial, viral, or other infection that is uncontrolled or requiring intravenous (IV) antimicrobials for management.
11. Uncontrolled or active infectious diseases, such as human immunodeficiency virus (HIV) infection, acute or chronic active hepatitis B or C, epstein-barr virus (EBV), and cytomegalovirus (CMV) infection.
12. History or presence of CNS disorder such as seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with CNS involvement.
13. Subjects with cardiac atrial or cardiac ventricular lymphoma involvement.
14. History of myocardial infarction, cardiac angioplasty or stenting, unstable angina, or other clinically significant cardiac disease within 12 months of enrollment.
15. Expected or possible requirement for urgent therapy within 6 weeks due to ongoing or impending oncologic emergency (eg, tumor mass effect, tumor lysis syndrome).
16. Primary immunodeficiency.
17. History of autoimmune disease (e.g. Crohn's, rheumatoid arthritis, systemic lupus) resulting in end organ injury or requiring systemic immunosuppression/systemic disease modifying agents within the last 2 years.
18. History of symptomatic deep vein thrombosis or pulmonary embolism requiring systemic anticoagulation within 6 months of enrollment.
19. Any medical condition likely to interfere with assessment of safety or efficacy of study treatment.
20. History of severe immediate hypersensitivity reaction to any of the agents used in this study.
21. Vaccine ≤ 6 weeks prior to planned start of conditioning regimen.
22. In the investigator's judgment, the subject is unlikely to complete all protocol-required study visits or procedures, including follow-up visits, or comply with the study requirements for participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2026-04-25 (Estimated); Study Completion 2027-04-25 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Incidence of adverse events (AEs) defined as DLT | First infusion date of CAR-T cells up to 28 days
  DLT is defined as any AE related to the investigational drug that occurs within 28 days after administration of the ATHENA-2 CAR-T and meets any one of the criteria listed in the DLT criteria. The severity of AE will be assessed according to NCI-CTCAE v5.0. Cytokine release syndrome (CRS) and immune cell-associated neurotoxicity syndrome (ICANS) will be evaluated according to the standards released by ASTCT in 2019. GvHD according to criteria defined by the Mount Sinai Acute GVHD International Consortium.
  * Grade 3 acute GVHD (aGVHD) that is not resolved to Grade 1 or 2 within 7 days, with the exception of isolated skin involvement aGVHD;
  * Grade 4 CRS or grade 3 CRS that is not resolved to grade 2 or lower within 2 weeks;
  * Grade 3 ICANS lasting for ≥7 days or Grade 4 ICANS;
  * Any other Grade ≥4 and Grade 3 AEs related to the ATHENA-2 CAR-T that lasts for ≥14 days, except hematology toxicity.
Phase 1: Recommended phase 2 dose (RP2D) | 12 months
  The RP2D will be determined based on the maximum tolerated dose, occurrence of dose-limiting toxicity, the obtained efficacy results, pharmacokinetics/pharmacodynamics and other data according to the phase 1.
Phase 2: 3-month objective response rate (ORR) | 3 months
  ORR is defined as the proportion of patients who have achieved complete response (CR) and partial response (PR) assessed by investigators.
Phase 2: Complete response (CR) rate | 24 months
  CR is assessed by investigators and based on the Lugano 2014 assessment criterion. CR rate is defined as the proportion of patients who have achieved CR assessed by investigators.
Phase 2: Duration of Response (DOR) | 24 months
  DOR is defined as the date of their first CR or PR (which is subsequently confirmed) to PD assessed by investigators, or death regardless of cause.
Phase 2: Overall Survival (OS) | 24 months
  OS is defined as the time from CAR-T cells infusion to the date of death. Subjects who have not died by the analysis data cutoff date will be censored at their last contact date.
Phase 2: Progression Free Survival (PFS) | 24 months
  PFS is defined as the time from the CAR-T cells infusion date to the date of disease progression assessed by investigators, or death any cause. Participants not meeting the criteria for progression by the analysis data cutoff date were censored at their last evaluable disease assessment date.

SECONDARY OUTCOMES:
Phase 1 and phase 2: Pharmacokinetics: Level of ATHENA-2 CAR-positive T cells circulating in blood over time | 12 months
  The absolute count of ATHENA CAR-T cells in peripheral blood is assessed by flow cytometry. Blood samples were collected before and one year after cell infusion (until CAR-T cells were not detected for two consecutive times) to detect the number and copy number of CAR-T cells, and to evaluate the pharmacokinetics of CAR-T.
Phase 1 and phase 2: Pharmacodynamics: Level of CD19+ cells in peripheral blood | 12 months
  The level of CD19+ cells in peripheral blood will be detected by flow cytometry.
Phase 1 and phase 2: Level of serum cytokines in peripheral blood | Up to 28 days after infusion
  The level of serum cytokines in peripheral blood will be detected by enzyme-linked immuno sorbent assay.
Phase 1: 3-month ORR | 3 months
  ORR is defined as the proportion of patients who have achieved CR and PR assessed by investigators and based on the Lugano 2014 assessment criterion.
Phase 1: OS | 24 months
  The definition of OS has already been mentioned above.
Phase 1: PFS | 24 months
  The definition of PFS has already been mentioned above.
Phase 2: Incidence of AEs | 24 months
  AEs are defined as any adverse medical event from the date of enrollment to 24 months after CAR-T cells infusion.

OTHER OUTCOMES:
Phase 1: Level of donor-specific antibody (DSA) in blood. | 12 months
  DSA refers to the specific antibody produced in the recipient's body targeting donor antigens after receiving CAR-T cell infusion from healthy donors.
Phase 1: Level of human anti-mouse antibodies (HAMA) | 12 months
  The level of human against murine scFv antibodies in blood.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Biotherapeutic Department of Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Biotherapeutic Department of Chinese PLA General Hospital, Beijing
  - School of Life Sciences, Peking University, Beijing

IPD SHARING:
Plan to Share IPD: No